CLINICAL TRIAL: NCT02173197
Title: Study on the Effectiveness of Occupational Therapy Intervention in Complex Patients.
Brief Title: Effectiveness of Occupational Therapy Intervention in Complex Patients
Acronym: OT
Status: Completed | Type: Observational
Sponsor: Stefania Costi (Other)
Collaborators: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor-Investigator, Stefania Costi, Physical Therapist, University of Modena and Reggio Emilia
Organization: University of Modena and Reggio Emilia (Other)
Other Study IDs: TO_Pilota
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Complex Patients: Patients With High Level of Complexity Regardless of the Pathology of Origin
Keywords: Occupational Therapy; Complex patients; Occupational performance problem; Rehabilitation Complexity Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OT arm: Through the initial evaluation of the complex patients' needs, the OT will propose a targeted intervention to the needs emerged and decide which approach will use to achieve the goal (i.e. compensatory or restorative).
  We will describe the characteristics of the population included and identify common needs and problems of the complex patients through the COPM.
  The needs and problems identified will be grouped into macro-areas, and the OT will propose the appropriate treatment on the basis of the area identified, the patient's needs and the available resources regardless of the origin of the disease.

SUMMARY:
To date, there are no studies that demonstrate that the intervention of Occupational Therapy (OT) in patients considered to be complex, regardless of diagnosis, could improve clinical and functional outcome for the patient.

For this reason, we intend to undertake a study that will allow us to deepen the knowledge about the impact of the OT on in-hospital patients considered "complex" according to the assessment by the Rehabilitation Complexity Scale (RCS ).

Our hypothesis is that the intervention of OT can improve their care by qualified and focused on the needs of the person interventions.

DETAILED DESCRIPTION:
We will therefore first af all to implement an observational pilot study, aimed at defining the characteristics and needs of the population in question, and the OT intervention "protocol". This information will then be used to implement a subsequent randomized controlled trial designed to demonstrate the effectiveness of the OT intervention on the basis of clinically relevant outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* in charge of the rehabilitation ward of the hospital
* defined complexes as assessed by RCS
* consent to the processing of sensitive data for research purposes.

Exclusion Criteria:

* primary psychiatric conditions
* language barrier;
* cognitive impairment
* communicative disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-hospital complexes patients as defined by way of the Rehabilitation Complexity Scale, regardless of the diagnosis and in charge of the rehabilitation ward
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | enrollment
  Canadian occupational performance measure

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Fugazzaro, MD, Principal Investigator — Azienda USL Reggio Emilia - IRCCS; Claudio Tedeschi, MD, Study Chair — Arcospedale Santa Maria Nuova - IRCCS

REFERENCES:
- [Result] Schiavi M, Costi S, Pellegrini M, Formisano D, Borghi S, Fugazzaro S. Occupational therapy for complex inpatients with stroke: identification of occupational needs in post-acute rehabilitation setting. Disabil Rehabil. 2018 May;40(9):1026-1032. doi: 10.1080/09638288.2017.1283449. Epub 2017 Feb 7. PMID 28264614